CLINICAL TRIAL: NCT05487144
Title: Self-management EdUcation and SuPport to Promote PsychOsocial Health Among StRoke Survivors and Informal Caregivers in a VirTual Stroke Community (SUPPORT): A Pilot Project
Brief Title: Self-management EdUcation and SuPport to Promote PsychOsocial Health Among StRoke Survivors and Informal Caregivers in a VirTual Stroke Community (SUPPORT)
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jennifer Beauchamp, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-SN-21-1005
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Stroke
Keywords: depression; anxiety
MeSH Terms: conditions — Stroke; Depression; Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Behavioral: Learning in a Virtual Environment (LIVE)

INTERVENTIONS:
Behavioral: Learning in a Virtual Environment (LIVE) — Phase 1 of the study will be a one-time meeting, either remote or in-person to complete V.E. training and fill out questionnaires. Phase 2 of the study is the 8 week intervention implementation.Participants will access the V.E. community from their homes on a computer with broadband internet. During the first four weeks of the intervention, participants will be required to come into the V.E. at least once per week for at least one hour. For the last four weeks, V.E. participation is strongly encouraged, but not required. The content in the V.E. will focus on psychosocial health and stroke recovery, and the messaging in the VE will be updated bi-weekly to encourage retention and engagement. Group meetings led by the study PI, a psychologist, or another trained member of the research team at least once a week will be offered. During the intervention period, VE-specific data will be collected continuously. Phase 3, will include a survey and a focus group interview via online platform.

SUMMARY:
The purpose of this study is to create a virtual stroke community for stroke survivors and informal caregivers of stroke survivors by customizing an existing VE intervention to incorporate real-time, stroke-specific, psychosocial self management education (SME) and social interactions, to test feasibility, acceptability, and usability of the customized intervention for stroke survivors and informal caregivers of stroke survivors and to obtain and explore data to derive evidence-based hypotheses and properly design and conduct a future, larger trial to demonstrate treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors that have experienced an ischemic or hemorrhagic stroke event and their caregivers
* can read, write, and speak English
* are able to provide written consent
* are computer literate (have used a computer for ≥1 month)
* have access to a computer with broadband internet at home
* understand how to use the Internet (accessed the Internet on ≥2 occasions)

Exclusion Criteria:

* reside outside of the home
* Montreal Cognitive Assessment score of <9 indicating moderate to severe impairment
* Caregivers that provide long-distance care. I

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by the number of participants enrolled in the study | post intervention (8 weeks from baseline of last participant )
  This will be defined as the number enrolled divided by the number of eligible individuals screened
Feasibility as assessed by the number of participants who complete the study | post intervention (8 weeks from baseline of last participant )
Feasibility as assessed by the number of participants who complete the data collection forms | post intervention (8 weeks from baseline of last participant )
Usability as assessed by the perceived usefulness score | post intervention (8 weeks from baseline)
Usability as assessed by the perceived ease of use scores | post intervention (8 weeks from baseline)
  This has 10 items, each scored form 1(strongly disagree) to 5(strongly agree), higher score meaning higher perceived ease of use
Usability as assessed by the number of times the participants log in | post intervention (8 weeks from baseline)
Usability as assessed by the time spent in the environment in minutes | post intervention (8 weeks from baseline)
Acceptability as assessed by the number of VE Meetings attended | post intervention (8 weeks from baseline)
Acceptability as assessed by the number of VE objects manipulated | post intervention (8 weeks form baseline)
  Objects manipulated are the resources interacted with

SECONDARY OUTCOMES:
Change in perceived social support as assessed by the Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline, post intervention (8 weeks after baseline)
  This is a 12 item scale , each question is scored from 1(very strongly disagree) to 7(very strongly agree) for a maximum score of score of 84, a higher number indicating more social support
Change in post stroke depression as assessed by the Patient Health Questionnaire-9 score (PHQ-9) | Baseline, post intervention (8 weeks after baseline)
  This is a 9 item questionnaire, each scored from 0(not at all) to 3(nearly every day), a higher number indication g more depression
Change in anxiety as assessed by the Generalized Anxiety Disorder-7 score | Baseline, post intervention (8 weeks after baseline)
  This is a 7 item questionnaire, each is scored from 0(not at all) to 3(nearly every day) a higher number indicating more anxiety
Change in loneliness as assessed by the UCLA loneliness scale scores | Baseline, post intervention (8 weeks after baseline)
  This is a 20 item questionnaire, each one is scored form 1(never) to 4(always). Scores for questions 1,5,6,9,10,15,16,19 and 20 are reversed(i.e. 1=4,2=3,3=2,4=1)and the scores for each item is then summed together, higher number indicating more loneliness
Change in caregiver burden as assessed by the Zarit Burden Interview (ZBI) | Baseline, post intervention (8 weeks after baseline)
  This is a 22 item questionnaire,each one scored from 0(never)-4(nearly always) higher core indicating more burden
Change in self efficacy ( ability to perform tasks or behaviors) as assessed by the PROMIS General Self-efficacy Form | Baseline, post intervention (8 weeks after baseline)
  This is a 10 item questionnaire, each one is scored from 1(not at all true) to 4(exactly true), a higher number indicating a better outcome
Change in emotional support as assessed by the NIH Emotional Support Form | Baseline, post intervention (8 weeks after baseline)
  This is an 8 item questionnaire, and each is scored form 1(never)-5(always), for a maximum score of 40, a higher number indicating higher levels of emotional support
Change in instrumental support as assessed by the PROMIS Short Form v2.0 | Baseline, post intervention (8 weeks after baseline)
  This is an 8 item questionnaire, and each is scored form 1(never)-5(always), for a maximum score of 40, a higher number indicating higher levels of instrumental support
Change in ability to recover form stress as measured by the Brief Resilience Scale | Baseline, post intervention (8 weeks after baseline)
  This is a 6 item questionnaire scored from 1 (strongly disagree) to 5 (strongly agree) a higher number indicating a better outcome?
Change in the amount that pain interferes with daily life as assessed by the PROMIS Short Form Pain Interference v 1.0 8a | Baseline, post intervention (8 weeks after baseline)
  This is an 8 item questionnaire and each is scored from 1 (not at all) to 5 (very much) a higher number indicating a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Beauchamp, PhD, RN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beauchamp JES, Wang M, Leon Novelo LG, Cox C, Meyer T, Fagundes C, Savitz SI, Sharrief A, Dishman D, Johnson C. Feasibility and user-experience of a virtual environment for social connection and education after stroke: A pilot study. J Stroke Cerebrovasc Dis. 2024 Feb;33(2):107515. doi: 10.1016/j.jstrokecerebrovasdis.2023.107515. Epub 2023 Dec 7. PMID 38064972